CLINICAL TRIAL: NCT06537219
Title: Thoracolumbar Fascia Stiffness and Pain Parameters
Brief Title: Changes in Thoracolumbar Fascia Stiffness and Pain Parameters in Young Patients With Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, NAİME ULUG, Assistant Professor, Atılım University
Other Study IDs: E-59394181-604.01-79246
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Pain; Back Pain; Fascia
Keywords: non-spesific back pain; thoracolumbar fascia; stiffness; pain thresold
MeSH Terms: conditions — Pain; Back Pain | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- back pain group: participants with chronic back pain( pain duration at least 3 months) aged between 18 and 50 years , male and female participanst will be included in the study. Those with orthopaedic, neurological and systemic diseases will be excluded from the study.
  Interventions: Other: Assessment
- control group: healty male and female participants aged between 18 and 50 years
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment of pain severity,pain thresold of the fascia, pain sensitivity

SUMMARY:
This study aims to investigate the biomechanical parameters of thoracolumbar fascia (TLF) and pain-related properties including pain intensity, pressure pain threshold (ppt) and pain sensitivity in young adults with non-specific chronic low back pain (LBP), both those experiencing chronic low back pain (LBP) and without LBP.

DETAILED DESCRIPTION:
Non-specific low back pain has become a serious public health problem in latest years. The prevalence of low back pain is reported to be 84% in lifetime (1). Recently, an increasing number of studies have reported that fascia, due to its rich nociceptive innervations, may play a role in chronic pain, especially in some non-specific low back pain conditions .

This study will conducted with a total of 50 participant, including those with chronic lower back pain in the experimental group and the control group.

Both groups underwent assessments related to pain properties. Specifically, the Numerical Pain Scale(NMS) will be used to assess subjective pain intensity(4), the Digital Algometer for assessing pressure pain treshold(5), the Pain Sensitivity Scale(PSS) pain sensitivity(6) and the Myotonometer MyotonPRO biomechanical parameters, including stiffness(s), elasticity(d) and tonus (f) of the TFL at the level of Lumbal 1,3 vertebrae(L1,L3) and under 12th costa (7-10). SPSS 23.0 will be used for statistical analysis. p<0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* chronic back pain participants more than 3 months

Exclusion Criteria:

* Those with orthopaedic, neurological and systemic diseases will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Academic staff and university students at Atılım University will constitude the study population.
  Sample size is calculated with 85% power. 50 participants( 25 experiment,25 control group) will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Scale(NMS | 1 month
  pain assessment
Fascia stiffness | 1month
  thoracolumbar fascia stiffness assessment
the Pain Sensitivity Scale(PSS) | month
  Pain sensitivity assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No